CLINICAL TRIAL: NCT02542397
Title: LCI-NOS-PAIN-001: A Prospective, Pharmacogenomic-Driven Pilot Study of Pain Management in Oncology Outpatients
Brief Title: LCI-NOS-PAIN-001: A Prospective, Pharmacogenomic-Driven Study of Pain Management in Oncology Outpatients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early study closure due to limited internal resources to continue enrollment.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LCI-NOS-PAIN-001
Record Dates: First submitted 2015-09-02; First posted 2015-09-07 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2021-03

CONDITIONS: Malignant Tumor of Ill-defined Site
MeSH Terms: interventions — Pharmacogenomic Testing

STUDY DESIGN:
Intervention Model Description: Enrolled subjects all receive pharmacogenomic testing with the intention of guiding pain management. This single-arm trial is testing against a published historical control.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pharmacogenomic Testing (Experimental): Pharmacogenomic test results to guide drug/dose modifications
  Interventions: Genetic: Pharmacogenomic Testing

INTERVENTIONS:
Genetic: Pharmacogenomic Testing — Pharmacogenomic test results to guide drug/dose modifications

SUMMARY:
About half of all cancer patients seen in oncology clinics have pain at initial assessment; pain relief within a one-month period is seen in approximately one third of these patients and pain worsening in about one fifth. Risk factors for under-treatment of cancer pain include age older than 65 years, minority status, and inadequate pain assessment practices. There is a need for better methods of opioid drug/dose selection and identification of risk factors for worsening pain. Pharmacogenomic approaches offer insight into the genetic variables that impact the pharmacokinetic and pharmacodynamic behavior of opioids. Translating pharmacogenomic results into actionable prescribing decisions may ultimately enable a personalized approach to pain management, increasing the chance of significant pain improvement. Cancer outpatients with uncontrolled malignant pain will be offered a pharmacogenomic test through participation in the study. The results of this test will be used to modify their pain regimen, if applicable.

DETAILED DESCRIPTION:
All subjects will be assessed and prescribed a pain regimen as part of standard practice at the initial visit. Subjects will provide a buccal swab for pharmacogenomic testing and will be discharged on their initial pain regimen.

After the initial visit, subjects will be asked to rate their daily pain on a scale of 0-10. A coordinator will follow up with the subject within 7 days (Assessment #1). Subjects will be asked to report information about their pain scores, pain medication use, and caffeine intake, in addition to any bothersome symptoms. Subjects who continue to have "uncontrolled pain", are experiencing bothersome symptoms, and/or requests for a drug/dose modification will have his/her drug/dose modified using the pharmacogenomic test results. If the subject has had significant pain improvement, stable mild pain and/or is satisfied with their level of pain at the assessment (regardless of pain score), he/she will be recommended to continue the current drug/dose and return to clinic on day 30 for the final follow-up. Subjects will be told to call if their pain becomes intolerable or if they experience bothersome symptoms after Assessment #1 for further drug/dose modification if needed prior to day 30.

The coordinator will follow up with the subjects receiving a drug/dose modification after another 7 days (Assessment #2). Subjects who have now had significant pain improvement, stable mild pain, and/or are satisfied with their level pain at the assessment (regardless of pain score) will continue on the same regimen. If the subjects' pain is still "uncontrolled", they are experiencing bothersome symptoms, and/or they request a drug/dose modification, their drug/dose will be modified accordingly. Subjects will be told to call if needed, otherwise they will be seen in clinic on day 30 (Final Assessment).

If the subject experiences intolerable pain prior to any scheduled assessment, the subject will call for appropriate drug/dose modification.

ELIGIBILITY:
Inclusion Criteria:

* Presence of uncontrolled malignant pain (score of greater than or equal to 2 on an 11 point scale [0-10]) as diagnosed and assessed by the Investigator, using the Edmonton Symptom Assessment Scale (ESAS).
* Documentation of any stage of cancer of any tumor location (solid or hematological).
* At least 18 years of age.
* Either nociceptive or neuropathic pain.
* Able to understand and be willing to sign the study consent form.

Exclusion Criteria:

* Inpatient service at baseline visit.
* Significant dysphagia and inability to swallow oral medications as determined by the Investigator.
* Active or recent (within one year) drug and/or alcohol abuse as determined by the Investigator.
* Significant baseline cognitive impairment, as determined by the Investigator. Known (anaphylactic) hypersensitivity to any opioid.
* Severe oral mucositis that would impair proper buccal testing as determined by the Investigator.
* Receiving concurrent rehabilitation medicine care, nociception modulation (e.g., electrical stimulation), use of modalities with physiologic effects that indirectly influence nociception (e.g., light, laser therapy), or any other non-pharmacologic approaches to pain management other than exercise, rest, ice, compression, and elevation (RICE).
* Presence of major psychiatric disorders as determined by the Investigator.
* Receiving active treatment or prophylaxis for epilepsy.
* Unable or unwilling to sign the study consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-09; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jai Patel, PharmD, Principal Investigator — Atrium Health Levine Cancer Institute
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

REFERENCES:
- [Derived] Patel JN, Boselli D, Symanowski J, Wodarski S, Turner S, Slaughter C, Myers M, Edwards R, Susi B, Greiner R, Edelen C. Pilot study of multi-gene pharmacogenetic testing for pain management in oncology palliative medicine. Pharmacogenomics. 2021 Aug;22(12):737-748. doi: 10.2217/pgs-2021-0037. Epub 2021 Aug 20. PMID 34414777

RESULTS

PARTICIPANT FLOW:
Groups:
- Pharmacogenomic Testing: Cancer outpatients with uncontrolled malignant pain undergo a pharmacogenomic panel (by buccal swab) with the intent of informing pain management.
Period: Overall Study
Arm/Group | Pharmacogenomic Testing
Started | 75 (75 subjects were enrolled to the study (i.e., submitted buccal swab).)
Completed | 59 (54 enrolled subjects provided pain scores at baseline and final assessments within 30 +/- 7 days.)
Not Completed | 16
Not completed — Death | 2
Not completed — Physician Decision | 6
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: The baseline analysis population is defined as all enrolled subjects (i.e., submitted buccal swab for pharmacogenomic testing).
Arm/Group | Pharmacogenomic Testing
Number analyzed (Participants) | 75
Age, Continuous [Median (Full Range); unit: years] | 61 [30 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 58
  More than one race | 0
  Unknown or Not Reported | 1
Cancer type [Count of Participants; unit: Participants]
  Breast | 14
  Gastrointestinal | 12
  Gynecologic | 8
  Multiple Myeloma | 11
  Thoracic | 10
  Genitourinary | 5
  Cutaneous malignancies | 6
  Other | 9
Stage of cancer (as captured from the Medical Record and determined by the TNM system of the AJCC) [Count of Participants; unit: Participants]
  1 or 2 | 13
  3 or 4 | 57
  Other | 5

OUTCOME MEASURES:

1. Primary Outcome: Rate of Pain Improvement as Measured Using the Edmonton Symptom Assessment Scale (ESAS) From Baseline Assessment (Day 0) to Final Assessment on Day 30 +/- 7
Description: Proportion of subjects achieving significant pain improvement over a one month period (30 days +/- 7) (defined as a ≥ 2 point decrease from baseline pain score on an 11-point scale [0-10]) in oncology outpatients receiving pharmacogenomic testing.
Time Frame: Enrollment to Final Assessment (30 +/- 7 days from Baseline Assessment (Day 0))
Population: The evaluable population is defined as those enrolled subjects providing pain scores at Baseline Assessment (Day 0) and Final Assessment (Day 30 +/- 7).
Measure: Number (95% Confidence Interval); unit: proportion of evaluable participants
Groups:
- Pharmacogenomic Testing: Evaluable Population: Enrolled subjects providing pain scores at Baseline Assessment (Day 0) and Final Assessment (Day 30 +/- 7).
Arm/Group | Pharmacogenomic Testing: Evaluable Population
Number analyzed (Participants) | 54
proportion of evaluable participants | .5556 [.4140 to .6908]
Statistical Analysis 1: Comparison: Pharmacogenomic Testing: Evaluable Population; A single-stage design was used to test the hypothesis that the pain improvement rate, assessed by the Edmonton Symptom Assessment Scale, is <= 0.30. Our study targeted enrollment of 71 evaluable subjects for the final analysis; 54 subjects met the criteria at study closure. Assuming a one-sided alpha=0.10 significance level, 71 evaluable subjects would provide approximately 90% power to reject the null hypothesis (based on an exact binomial test) assuming the true pain improvement rate is 0.45; Test type: Superiority — It has been reported that, based on the Edmonton Symptom Assessment Scale (ESAS) pain scale, about 30% of cancer patients receiving standard of care pain management experienced >= 2-point improvement in pain score between visits [Ref]. Ref: Scharpf, J., et al., The role of pain in head and neck cancer recurrence and survivorship. Arch Otolaryngol Head Neck Surg, 2009. 135(8): p. 789-94; p < 0.0001, Exact binomial test of proportions — The a priori threshold for statistical significance was alpha = 0.10; Exact binomial proportion = .5556, 95% CI 2-sided [.4140 to .6908]

2. Secondary Outcome: Morphine Equivalent Daily Doses (MEDD) in Milligrams
Description: Describe the distribution of morphine equivalent daily dose (MEDD) in the evaluable population. The MEDD was calculated and recorded at the Final Assessment for each subject by converting the subject's total daily opioid consumption at the Final Assessment to morphine equivalent doses using the following website: http://www.globalrph.com/narcoticonv.htm (widely used across many health systems for drug/dose conversions and fully referenced).
Time Frame: Final Assessment (30 +/- 7 days from Baseline Assessment (Day 0))
Population: as for outcome 1
Measure: Median (Full Range); unit: milligrams
Groups:
- Pharmacogenomic Testing: Evaluable Population: Enrolled subjects providing pain scores at baseline assessment and a final assessment within 30 +/- 7 days.
Arm/Group | Pharmacogenomic Testing: Evaluable Population
Number analyzed (Participants) | 54
milligrams | 90 [0 to 789]

3. Secondary Outcome: Percentage of Subjects With an Actionable Genotype, Defined as the Presence of Any Mutation(s) That is (Are) Used to Guide a Drug/Dose Modification
Description: An actionable genotype is defined as the presence of at least one mutation that is used to guide a drug/dose modification during Assessment 1, Assessment 2, or any unscheduled visit.
Time Frame: Enrollment to Final Assessment (30 +/- 7 days from Baseline Assessment (Day 0))
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of evaluable participants
Arm/Group | Pharmacogenomic Testing: Evaluable Population
Number analyzed (Participants) | 54
percentage of evaluable participants | 33.33 [21.09 to 47.47]

ADVERSE EVENTS:
Time Frame: From enrollment date (i.e., buccal swab is collected) (Day 0) to the final study assessment on Day 30 +/- 7.
Description: Opioid-related adverse events were summarized and attributed based on Common Terminology Criteria for Adverse Events version 4.03. Adverse events deemed "possibly", "probably", and "definitely related" to opioid use by the Investigator were summarized for the study.
Arm/Group | Pharmacogenomic Testing
All-Cause Mortality (participants affected / at risk) | 2/75
Serious Adverse Events (participants affected / at risk) | 2/75
Other Adverse Events (participants affected / at risk) | 34/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pharmacogenomic Testing (N=75)
Death NOS (General disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pharmacogenomic Testing (N=75)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (3)
Confusion (Psychiatric disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 7 (8)
Delirium (Psychiatric disorders) | 2 (2)
Dizziness (Nervous system disorders) | 6 (6)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Fatigue (General disorders) | 7 (9)
Gait disturbance (General disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions - Other, Weakness in joints (General disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (3)
Hypersomnia (Nervous system disorders) | 1 (1)
Injury, poisoning and procedural complications - Other, Chin laceration (Injury, poisoning and procedural complications) | 1 (1)
Nausea (Gastrointestinal disorders) | 13 (14)
Nervous system disorders - Other, Change in mental status (Nervous system disorders) | 2 (2)
Neuralgia (Nervous system disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2)
Somnolence (Nervous system disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
Early study closure due to limited internal resources to continue enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-07-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT02542397/Prot_SAP_000.pdf
  • Informed Consent Form (2015-12-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT02542397/ICF_001.pdf